CLINICAL TRIAL: NCT00663221
Title: Study of the Osteoprotector Effects of a Milk Product Based on Anthocyans and Enriched in Calcium and Vitamin D
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Elvir SAS (Industry)
Collaborators: University Hospital, Clermont-Ferrand (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: LC2 Atlas
Record Dates: First submitted 2008-04-14; First posted 2008-04-22 (Estimated); Last update posted 2009-07-07 (Estimated); Status verified 2009-07

CONDITIONS: Osteoporosis
Keywords: Osteoporosis prevention
MeSH Terms: conditions — Osteoporosis | interventions — Calcium; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- 1 (Placebo Comparator)
  Interventions: Dietary Supplement: placebo
- 2 (Experimental)
  Interventions: Dietary Supplement: Anthocyans, Calcium and Vitamin D

INTERVENTIONS:
Dietary Supplement: Anthocyans, Calcium and Vitamin D
  Arms: 2
Dietary Supplement: placebo
  Arms: 1

SUMMARY:
We hypothesize that anthocyans with calcium and vitamin D have a positive effect on bone reshaping in menopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Aged between 50 and 65 years
* Between 1 and 5 years menopause
* IMC between 19 and 30 kg/m²

Exclusion Criteria:

* Medical Treatment for bone metabolism
* Vitamin D not including in the range of 20nmoles<25(OH)<100nmoles/l
* Vegan and vegetarian diet
* Regular consumption of food supplementary benefits
* Lactose intolerance
* While dieting

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2008-03

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France